CLINICAL TRIAL: NCT02225743
Title: Observational Examination of Thermoregulation in Total Joint Arthroplasty
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Other Study IDs: Thermoregulation Total Joint; Pro00035290 (Other: MUSC)
Record Dates: First submitted 2014-08-21; First posted 2014-08-26 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Hypothermia
Keywords: Hypothermia; Total Hip Joint Prosthesis; Total Knee Joint Prosthesis
MeSH Terms: conditions — Hypothermia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Joint Arthroplasty: Participants undergoing joint replacement
  Interventions: Other: Observation Of Temperature

INTERVENTIONS:
Other: Observation Of Temperature — Participants temperature will be recorded perioperatively.

SUMMARY:
Total joint patients have poor outcomes with infection since they are having permanent hardware implanted. Infection prevention in this group is therefore critical and a major source of discussion in both the orthopedic and anesthesia literature.

Hypothermia has been shown to increase the risk of infection and blood loss. However, studies have not examined when in the operation or how fast patients temperatures drop. This study will observe how patients' temperatures change during total joint arthroplasty. By identifying when body temperature changes occur, prevention strategies may be developed and implemented.

DETAILED DESCRIPTION:
Peri-operative hypothermia can have deleterious effects. While there is no standard consistent definition within the literature mild hypothermia is commonly defined as a core temperature between 34 and 36 °C. Mild hypothermia has been shown to increase the occurrence of surgical site infections, cardiac morbidity, coagulopathy leading to increased blood loss and transfusion requirements, impaired drug metabolism, and prolonged emergence from anesthesia. In addition, there is evidence that maintaining intra-operative normothermia can shorten hospital length of stay. Despite the fact that intra-operative temperature monitoring and warming are considered standard of care, peri-operative hypothermia in total joint arthroplasty patients remains an issue for several reasons. A large proportion of patient undergoing joint replacement are elderly, making them susceptible to peri-operative hypothermia. In addition, regional anesthesia causes vasodilation and promotes heat flow from the core to the periphery and impairs central and autonomic thermoregulation such that patients receiving neuraxial anesthesia can be particularly susceptible to perioperative hypothermia. Finally, core temperature monitoring is typically not used during regional anesthesia and hypothermia may go undetected for long periods of time.

The primary goal of this study was to examine the incidence of hypothermia during lower extremity arthroplasty. A secondary aim was to identify patient and operative factors associated with hypothermia in order to improve future preventative strategies. Our hypothesis was that peri-operative hypothermia occurs in the majority of patients undergoing lower extremity arthroplasty. In addition, we hypothesized that certain patient and anesthetic factors (such as low body mass index and receiving general anesthesia) would increase the incidence of hypothermia.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age and over that are scheduled to undergo total hip or total knee joint arthroplasty.

Exclusion Criteria:

* Patients unable to give informed consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 years or older that are having a total joint replacement surgery.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2014-08; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia H Wilson, MD, Principal Investigator — Medical University of South Carolina; Wanda Jones, Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Kurz A. Thermal care in the perioperative period. Best Pract Res Clin Anaesthesiol. 2008 Mar;22(1):39-62. doi: 10.1016/j.bpa.2007.10.004. PMID 18494388
- [Background] Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. Study of Wound Infection and Temperature Group. N Engl J Med. 1996 May 9;334(19):1209-15. doi: 10.1056/NEJM199605093341901. PMID 8606715
- [Background] Seamon MJ, Wobb J, Gaughan JP, Kulp H, Kamel I, Dempsey DT. The effects of intraoperative hypothermia on surgical site infection: an analysis of 524 trauma laparotomies. Ann Surg. 2012 Apr;255(4):789-95. doi: 10.1097/SLA.0b013e31824b7e35. PMID 22388109
- [Background] Sun Z, Honar H, Sessler DI, Dalton JE, Yang D, Panjasawatwong K, Deroee AF, Salmasi V, Saager L, Kurz A. Intraoperative core temperature patterns, transfusion requirement, and hospital duration in patients warmed with forced air. Anesthesiology. 2015 Feb;122(2):276-85. doi: 10.1097/ALN.0000000000000551. PMID 25603202

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Joint Arthroplasty
Started | 120
Completed | 102 (18 patients chose not to participate on the day of surgery.)
Not Completed | 18
Not completed — Withdrawal by Subject | 18

BASELINE CHARACTERISTICS:
Arm/Group | Joint Arthroplasty
Number analyzed (Participants) | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 38
Total Knee Arthroplasty [Count of Participants; unit: Participants] | 54

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Hypothermia
Description: The incidence of ever being hypothermic (temperature < 36.0 °C at one or more measurements) was the primary outcome. All temperatures were assessed with an Exergen temporal thermometer (precise to 0.1 °C). Each temporal measurement was taken and recorded three times for accuracy and the mean value utilized for data analysis at each time point. Temperatures were measured upon (1) leaving holding area; (2) operating room (OR) arrival; (3) after anesthetic induction; (4) upper body forced air warmer initiation (used for all patients); (5) incision; (6-8) every 30 minutes after incision; (9) leaving the OR; and (10) arrival to PACU. OR temperature and humidity were recorded throughout.
Time Frame: Starting with temperature measurement prior to leaving preoperative holding for OR and ending after temperature taken on arrival in recovery room
Population: Ever hypothermic (temperature <36.0 degrees C) during the perioperative period
Measure: Count of Participants; unit: Participants
Groups:
- Hypothermia: Hypothermia was defined as a temperature less than 36.0 °C. .
Arm/Group | Hypothermia
Number analyzed (Participants) | 102
Participants | 74

ADVERSE EVENTS:
Arm/Group | Joint Arthroplasty
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No